CLINICAL TRIAL: NCT01656980
Title: Phase 3 Study of Carmustine Sustained Release Implant (CASANT) to Treat Newly Diagnosed Malignant Glioma
Brief Title: Safety and Efficacy Study of Intracranially Implanted Carmustine to Treat Newly Diagnosed Malignant Glioma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Lanjin Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LJ-Glioma 3. 3.0 Version
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Glioblastoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carmustine Sustained Release Implant (Experimental): For subjects in this group, they will accept intracranially implanted carmustine intraoperatively.
  Interventions: Drug: Carmustine
- Tumor Resection Surgery (Sham Comparator): For subjects in this control group, they accept no implants while gliomas maximally be resected.
  Interventions: Procedure: tumor resection surgery

INTERVENTIONS:
Drug: Carmustine — As Experimental group, subjects will accept specified wafers of carmustine in the cavity while gliomas maximally be resected.
  Other Names: Trade name: CASANT; Other name: BCNU
  Arms: Carmustine Sustained Release Implant
Procedure: tumor resection surgery — For this group, subjects will accept routine tumor resection surgery and place no implant wafers.
  Other Names: blank control group
  Arms: Tumor Resection Surgery

SUMMARY:
The purpose of the study is to determine the safety and efficacy of intracranially implanted Carmustine in the treatment of patients with primary malignant glioma.

DETAILED DESCRIPTION:
Malignant gliomas recur mostly 2 cm within originated area. Local therapies therefore become particular important. Gliadel wafer developed in the States and marketed in the developed countries is an example of such treatments. The product in this study, Carmustine Sustained Release Implant (CASANT), is similar to that of Gliadel wafer as for the API(Active Pharmaceutical Ingredient), but different as for drug delivering system. As required, the preliminary clinical studies were conducted in China. Based on the results of phase I/II , 8-10 wafers containing given dose of BCNU will be administered intracranially in this phase III to the tumor resected cavity to investigate the safety and efficacy in the treatment of primary malignant glioma in 236 patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of high grade glioma(WHO III or above)by frozen or squash preparation;
* Patients must be 18 to 70 years old, signed ICF;
* At least 4 weeks after previous chemotherapy (6 weeks since nitrosoureas);
* KPS ≥ 60;
* Unilateral, Supratentorial, solitary lesion and not crossing the midline
* No obvious important organ dysfunction: Hepatic function:Serum total bilirubin ≤1.5 times upper limit of laboratory normal; Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT)<2.5 times upper limit of laboratory normal; Renal function:Serum creatinine ≤1.5 times upper limit of laboratory normal;
* Not Pregnant or lactating for women of childbearing potential.

Exclusion Criteria:

* Underwent cytoreductive surgery(excluded stereotactic biopsy);
* With chemotherapy or brain radiotherapy history;
* Tumor located at ventricular system, Open ventricle tumor cavity postoperatively;
* Concomitant with other life-threatening diseases and with life expectancy <12 months;
* Allergic to nitrosourea drugs;
* With history of intracranial radiotherapy or implant chemotherapy;
* With serious cardiac, pulmonary, hepatic and renal dysfunction, poor glycemic control;
* Experienced > 3 times of Large epilepsy within one month preoperatively.
* Investigators thought unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 15 months

SECONDARY OUTCOMES:
Progress Free Survival | 15 months
Overall Survival Rate at 12 months | 15 months
Karnofsky Performance Status(KPS) | 15 months
Quality of Life(QOL) | 15 months
Safety of intracranially implanted carmustine after maximal tumor resection | 15 months
  Occurrence rate of adverse event and serious adverse event revealed by laboratory test outcomes including blood routine and chemistry as well as physical examination, vital signs including blood pressure, temperature, respiratory rate , heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yan H Sun, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- See also: You will see subjects recruitment information when visiting above website. — http://lanjin.cn